CLINICAL TRIAL: NCT00989911
Title: Endothelin Blockade in Patients With Single Ventricle Physiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Jamil Aboulhosn, Assistant Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Actelion - 1
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Congenital Heart Disease
Keywords: Single ventricle congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosentan (Experimental): Bosentan
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — Bosentan 62.5 mg tablet taken orally twice daily for one month, followed by Bosentan 125 mg tablet taken orally twice daily for three months.
  Other Names: Tracleer

SUMMARY:
Recent studies have shown beneficial effects of sildenafil in patients with single ventricle congenital heart disease. The purpose of this study is to determine whether Bosentan, a drug with similar effects, will have similar benefit in this patient population.

DETAILED DESCRIPTION:
Patients enrolled in the study will take Bosentan. Baseline and follow up measurements will be collected then analyzed.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age
* Single ventricle congenital heart disease
* Require cardiac magnetic resonance imaging (MRI) for clinical purposes.

Exclusion Criteria:

* < 12 years of age
* Pregnancy or women who may become pregnant (sexually active and unwilling to use birth control)
* Patients taking cyclosporin or glyburide
* Patients with baseline liver dysfunction (aspartate aminotransferase or alanine aminotransferase > 3 times upper limit of normal)
* Contraindications to MRI (including pacemakers)
* Use of Bosentan within one month prior to enrollment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Aboulhosn, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Giardini A, Balducci A, Specchia S, Gargiulo G, Bonvicini M, Picchio FM. Effect of sildenafil on haemodynamic response to exercise and exercise capacity in Fontan patients. Eur Heart J. 2008 Jul;29(13):1681-7. doi: 10.1093/eurheartj/ehn215. Epub 2008 Jun 4. PMID 18534975
- [Background] Votava-Smith JK, Perens GS, Alejos JC. Bosentan for increased pulmonary vascular resistance in a patient with single ventricle physiology and a bidirectional Glenn shunt. Pediatr Cardiol. 2007 Jul-Aug;28(4):314-6. doi: 10.1007/s00246-007-0037-4. Epub 2007 Jun 11. PMID 17563825

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bosentan
Started | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Fontan, single ventricle patients all treated with Bosentan.
Arm/Group | Bosentan
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Blood Flow as Determined by MRI Velocity Encoding at 3-6 Months
Description: Magnetic resonance imaging-derived aortic flow
Time Frame: 3-6 months
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Bosentan
Number analyzed (Participants) | 7
L/min
  BaselineAortic Flow Volume | 3.3 (1.27)
  3-6 Month Aortic Flow Volume | 4.4 (0.9)
Statistical Analysis 1: Comparison: Bosentan; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Bosentan
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan (N=10)
fatigue (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No